CLINICAL TRIAL: NCT07162636
Title: FUNCTIONAL CAPACITY ANALYSIS THROUGH NEUROMUSCULAR ELECTRICAL STIMULATION COMBINED WITH RESISTANCE EXERCISE IN HOSPITALIZED SARCOPENIC INDIVIDUALS WITH ALCOHOLIC LIVER CIRRHOSIS: A DOUBLE-BLINDED RANDOMIZED CLINICAL TRIAL.
Brief Title: ELECTRICAL STIMULATION AND EXERCISE FOR MUSCLE LOSS IN CIRRHOSIS PATIENTS
Acronym: E-SEEM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitário Professor Edgard Santos (Other)
Responsible Party: Principal Investigator, Priscila Meireles Calil Fontana, Lead Investigator, M.S. in Rehabilitation Sciences., Hospital Universitário Professor Edgard Santos
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 88356025.7.0000.0049; 88356025.7.0000.0049 (Registry Identifier: Research Ethics Committee)
Record Dates: First submitted 2025-08-06; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-08

CONDITIONS: Sarcopenia; Liver Cirrhosis
Keywords: SARCOPENIA; LIVER CIRRHOSIS; NMES; HAND GRIP TEST; Five-Repetition Sit-to-Stand Test
MeSH Terms: conditions — Sarcopenia; Liver Cirrhosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NMES+ (Experimental): Participants will receive resistance exercise combined with NMES treatment.
  Interventions: Other: NMES -
- NMES - (Active Comparator): To treat and rehabilitate sarcopenia, participants will undergo physical therapy sessions using only resistance exercises
  Interventions: Other: NMES+

INTERVENTIONS:
Other: NMES+ — To treat and rehabilitate sarcopenia, participants will undergo physical therapy sessions, using resistance exercises combined with the use of NMES
  Arms: NMES -
Other: NMES - — To treat and rehabilitate sarcopenia, participants will undergo physical therapy sessions using only resistance exercises.
  Arms: NMES+

SUMMARY:
Introduction: Sarcopenia, whether primary or secondary, substantially impacts the quality of life of patients post-hospital discharge. Compromised functional capacity can lead to a high prevalence of readmissions. In this context, neuromuscular electrical stimulation (NMES), when combined with voluntary contraction (NMES+), emerges as a promising strategy for optimizing muscle strength gain.

Objective: To evaluate the efficacy of NMES+ in improving lower limb muscle strength and physical performance in hospitalized sarcopenic individuals with alcoholic cirrhosis.

Methods: This is a double-blind, randomized clinical trial. The Intervention Group will undergo NMES+, while the Control Group will perform resistance exercises. The sample will consist of individuals aged 47 to 70 years, diagnosed with sarcopenia through functional tests: handgrip strength and the 5-repetition sit-to-stand test. The protocol will be applied six times per week. Assessments will be conducted at hospital admission and discharge. Data will be analyzed using Student's T-tests for intergroup and intragroup comparisons; Spearman's or Pearson's correlation will assess the association between hospital readmission rates and physical function at hospital discharge. A p-value of 0.05 was set as statistically significant.

Expected Results: To observe a statistically significant increase in muscle strength and physical performance in the Intervention Group, and to find a negative correlation between improved physical function and hospital readmission rates.

Conclusion: This study is expected to contribute to more effective rehabilitation protocols, improving functionality and reducing hospital readmission in hospitalized patients with alcoholic liver cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized participants with alcoholic cirrhosis.

Exclusion Criteria:

* Five times sit-to-stand test (5xSTS) below the reference value according to the equation 5xSTS = 3.89 + (0.10 x age).
* Handgrip strength test (HGS) below 27Kgf for men and 16Kgf for women.

Ages: 47 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Efficacy of resistance exercise combined with NMES | 1 mounth
  The primary objective of this clinical trial is to increase muscle strength. This will be measured using the Handgrip Strength (HGS) test, a validated indicator that is particularly useful for hospitalized patients.

SECONDARY OUTCOMES:
Efficacy of resistance exercise combined with NMES | 1 month
  As a secondary objective, physical performance and functional lower limb strength will be evaluated, as they are directly impacted by sarcopenia. This assessment will be conducted using the five-repetition sit-to-stand test.
  Participants will be evaluated upon hospital admission and at discharge. A one-month post-discharge follow-up, conducted via telephone, will aim to monitor for potential hospital readmissions. This approach will allow for an investigation into the association between the readmission rate and physical function scores measured at the time of discharge.
  This study focuses on clinically relevant outcomes that directly impact patients' quality of life.

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF